CLINICAL TRIAL: NCT03273946
Title: Post-Marketing Observational Study to Evaluate Safety Profile of Flixotide 50 μg pMDI Treatment in Chinese Subjects With Asthma Aged 1-<4 Years
Brief Title: Post-marketing Safety Monitoring Program of Fluticasone Propionate (FP) in Chinese Subjects With Asthma Aged 1 to <4 Years
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 207734
Record Dates: First submitted 2017-09-05; First posted 2017-09-06 (Actual); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Asthma
Keywords: CCI18781; Observational; Post-marketing; Fluticasone propionate; Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects receiving fluticasone propionate: Eligible subjects will receive FP 50 µg twice daily inhaled via a pediatric pMDI with a face mask in clinical practice.
  Interventions: Drug: Fluticasone propionate

INTERVENTIONS:
Drug: Fluticasone propionate — Fluticasone propionate is an inhaled corticosteroid to be used via a pediatric spacer device with a face mask for prophylactic treatment of asthma.

SUMMARY:
For the prophylactic treatment of asthma, FP inhaled aerosol (Flixotide ®) administered via a pressurized metered-dose inhaler (pMDI) was approved in China in adults, adolescents older than 16 years of age and children aged 4 to 16 years. This post-marketing safety monitoring program will evaluate the safety profile of FP 50 micrograms (µg) inhaled via a pediatric spacer device with a face mask in Chinese subjects aged 1 to <4 years. The adverse drug reactions (ADRs) and predictors of these adverse reactions among subjects will be reported. This single arm observational study will include subjects prescribed with FP 50 µg inhaled via a pediatric spacer device with a face mask. The maximum duration of the study will be 12 weeks with 3 visits. Visit 1 (Day 1) will be on-site visit and will also mark the start of the observational program. The follow-up visits will be scheduled at Visit 2 (Week 4), and Visit 3 (Week 12) conducted on site or by telephone. A total of 150 asthmatic subjects who have been prescribed FP 50 µg treatment for appropriate medical use for the first time in China will be enrolled in the study. Flixotide is a registered trademark of GlaxoSmithKline (GSK) group of companies.

ELIGIBILITY:
Inclusion Criteria:

* An appropriately signed and dated assent must be obtained from the parent/guardian of the subject.
* Subjects with 1 to <4 years of age at Visit 1.
* Subjects who have been prescribed Flixotide 50 µg for a medically appropriate use for the first time will be included in this observational program; Flixotide 50 µg therapy should be in line with the approved dosing: 50 to100 µg twice daily; subjects should have the ability to inhale the doses via a pediatric spacer with a face mask appropriately; subjects who have been exposed to Flixotide 50 µg, 125 µg and 250 µg treatment previously will not be included.
* The parent/guardian of the subject must provide reliable contact information which includes home phone or cell phone for the follow up visits.
* The parent/guardian of the subject must have the ability to comply study procedures.
* Specific information regarding warnings, precautions, contraindications, AEs, and other pertinent information on Flixotide 50 μg that may impact subject eligibility is provided in the approved product label.

Exclusion Criteria:

-

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects aged between 1 to <4, diagnosed with asthma, who have been prescribed FP 50 µg for appropriate medical use for the first time in China will be included in this study.
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- China (2):
  - GSK Investigational Site, Shenzhen, Guangdong
  - GSK Investigational Site, Shanghai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single arm non-interventional, post-marketing safety monitoring study to evaluate safety of Chinese participants aged 1 to <4 years when using Flixotide 50 micrograms (μg) via a pediatric spacer device with a face mask in clinical practice. No medical intervention was received by participants during conduct of this study.
Pre-assignment Details: Total 158 participants were enrolled into this study. The study was conducted at 4 centers in China.
Groups:
- All Participants: The observational study included participants aged 1 to less than 4 years, who have been prescribed Flixotide 50 μg (recommended dosing 50 to 100 μg twice daily inhaled via a pediatric spacer device with a face mask) for appropriate medical use for the first time in clinical practice. The maximum study duration was 12 weeks with 3 visits. No medical intervention was received by participants during conduct of this study.
Period: Overall Study
Arm/Group | All Participants
Started | 158
Completed | 149
Not Completed | 9
Not completed — Withdrawal by Subject | 5
Not completed — Unwillingness of the guardian | 1
Not completed — Participant refused to use the drug | 2
Not completed — Participant relative refused to use drug | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 158
Age, Continuous [Mean (Standard Deviation); unit: Months] | 33.40 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 100
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Region of Enrollment is reported.
  Participants
    China: China | 158

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Adverse Drug Reaction (ADR)
Description: An AE is defined as any untoward medical event which occurred in a participant or clinical study participant, which is temporally associated with the use of the medical product, whether or not considered related to the product. An ADR is defined as AE related to study drug and listed in the package insert. Number of participants who had at least one AE or ADR are presented.
Time Frame: Up to Week 12
Population: Safety Analysis Population. It was defined as all the participants enrolled who received at least one dose of Flixotide 50 μg in clinical practice for appropriate medical use for the first time.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 158
Participants
  Any AE | 110
  Any ADR | 0

2. Primary Outcome: Number of Participants With Any Serious Adverse Event (SAE) or Non-SAE
Description: Any untoward medical occurrence resulting in death, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect, possible drug-induced liver injury or any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent serious outcomes were categorized as SAE. Number of participants who had at least one SAE or non-SAE are presented.
Time Frame: Up to Week 12
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 158
Participants
  Any non-SAE | 104
  Any SAE | 6

3. Primary Outcome: Number of Participants With Any New, Unexpected AE or Safety Signal
Description: An unexpected AE is defined as any adverse reaction whose nature and intensity have not been previously observed and documented for the study product (e.g. in the investigator brochure, product information). A safety signal is information on a new or known AE that may be caused by a medicine and requires further investigation. Number of participants with any new unexpected AE or safety signal are presented.
Time Frame: Up to Week 12
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 158
Participants
  Any unexpected AE | 0
  Any safety signal | 0

ADVERSE EVENTS:
Time Frame: In this non-interventional post-marketing safety monitoring study, non-SAEs and SAEs were collected up to Week 12 from start of the treatment in clinical practice. No medical intervention was received by participants during conduct of this study.
Description: Safety Analysis Population was used which included all participants enrolled who received at least one dose of Flixotide 50 μg in clinical practice for appropriate medical use for the first time.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/158
Serious Adverse Events (participants affected / at risk) | 6/158
Other Adverse Events (participants affected / at risk) | 104/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=158)
Pneumonia (Infections and infestations) | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=158)
Upper respiratory tract infection (Infections and infestations) | 47
Bronchitis (Infections and infestations) | 34
Rhinitis (Infections and infestations) | 9
Pharyngitis (Infections and infestations) | 8
Herpangina (Infections and infestations) | 8
Pneumonia (Infections and infestations) | 3
Rhinopharyngitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 4
Tonsillitis (Infections and infestations) | 4
Viral infection (Infections and infestations) | 4
Mycoplasma infection (Infections and infestations) | 3
Otitis media (Infections and infestations) | 2
Herpes pharyngitis (Infections and infestations) | 2
Molluscum contagious (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Pyrexia (General disorders) | 32
Influenza like illness (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Sensation of foreign body (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pain abdominal (Gastrointestinal disorders) | 1
Stomach inflammation (Gastrointestinal disorders) | 1
Indigestion (Gastrointestinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 4
Miliaria (Skin and subcutaneous tissue disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Urticarial rash (Skin and subcutaneous tissue disorders) | 1
Coughing (Respiratory, thoracic and mediastinal disorders) | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Balanoposthitis (Reproductive system and breast disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Abnormal hepatic function (Hepatobiliary disorders) | 1
Red blood cells urine (Investigations) | 1
Febrile convulsion (Nervous system disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT03273946/Prot_SAP_000.pdf